CLINICAL TRIAL: NCT04936906
Title: Patient Satisfaction Improvement and Quality of Life Measurement in Mohs Surgery
Brief Title: Mohs Surgery: Patient Satisfaction & Quality of Life (QOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180626
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra Care (EC) Treatment Group (Experimental): Participants in this group will receive the EC intervention pre and post standard of care (SoC) scheduled Mohs Surgery.
  Interventions: Behavioral: Extra Care (EC) Intervention
- Usual Care (UC) Group (Active Comparator): Participants in this group will receive the usual care provided to patients undergoing standard of care (SoC) scheduled Mohs Surgery.
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Behavioral: Extra Care (EC) Intervention — The EC intervention includes pre- and post- procedure calls from the surgeon, written educational material, personalized music during the operation, post-procedure skin cancer protection education, and are allowed to bring a guest into the procedure room.
  Arms: Extra Care (EC) Treatment Group
Other: Usual Care (UC) — Standard of care pre and post surgery management provided to patients undergoing Mohs Surgery.
  Arms: Usual Care (UC) Group

SUMMARY:
The purpose of this study is to examine whether there is significant difference between two groups: extra care (EC) and usual care (UC) in improvement of patients' quality-of-life (QoL) scores between the baseline and 90-day post-surgery in patients undergoing Mohs micrographic surgery (MMS).

ELIGIBILITY:
Inclusion Criteria:

1. Female and/or male subjects undergoing Mohs micrographic surgery for Basal Cell Carcinoma (BCC) and/or Squamous Cell Carcinoma (SCC).
2. Subjects must be at least 18 years of age.

Exclusion Criteria:

1. Subjects who are not able to complete the surveys (pre-surgery, 1 week post-surgery, and 3 months post- surgery)
2. Subjects under the age 18
3. Subjects unable to consent
4. Subjects who are not undergoing Mohs micrographic surgery for Basal Cell Carcinoma (BCC) or Squamous Cell Carcinoma (SCC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Change in PSQ Scores | Baseline, 3 months
  Patient Satisfaction Questionnaire (PSQ) is a 7 item questionnaire with a total score ranging from 7 to 35 with the higher score indicating greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No